CLINICAL TRIAL: NCT02686463
Title: Diagnosis and Treatment of Laparoscopy for Malignant Ovarian Cancer: an Open-label, Parallel, Randomized, Controlled Clinical Trial of Efficacy and Safety
Brief Title: Treatment for Malignant Ovarian Cancer: Laparoscopy vs Laparotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Qing Yang, Vice President, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QYang_001
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Ovarian Cancer
Keywords: malignant ovarian cancer; laparoscopy; laparotomy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- the laparoscopy group (Experimental): Patients who are randomized to the laparoscopy group.
  Interventions: Procedure: Laparoscopy
- the laparotomy group (Experimental): Patients who are randomized to the laparotomy group.
  Interventions: Procedure: Laparotomy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopy is an operation performed in the abdomen or pelvis through small incisions (usually 0.5-1.5 cm) with the aid of a camera. It can either be used to inspect and diagnose a condition or to perform surgery.
  Arms: the laparoscopy group
Procedure: Laparotomy — A laparotomy is a surgical procedure involving a large incision through the abdominal wall to gain access into the abdominal cavity. It is also known as a celiotomy.
  Arms: the laparotomy group

SUMMARY:
This trial is designed to compare diagnostic and therapeutic effects of laparoscopy vs. laparotomy on early malignant ovarian cancer, and to evaluate the efficacy and safety of laparoscopy in early malignant ovarian cancer.

DETAILED DESCRIPTION:
The principle for treating early-stage ovarian cancer is first to stage the cancer, and then to determine the optimal surgical and non-surgical treatments. Ovarian cancers mainly metastasize as extensive diffusions on surfaces of organs in the abdominal cavity. Although the most common ovarian cancer staging method is laparotomy, this procedure often misses upper abdominal metastases, especially on the diaphragm muscles, thus leading to inaccurate staging and prognostic assessments, and insufficient treatment.

A laparoscopic approach allows closer observation of relevant tissues, as these tissues are magnified in laparoscopies, which facilitates discovery of small lesions on surfaces of diaphragmatic muscle, liver and stomach fundus. Laparoscopes allow lavage of a wider area of the abdominal cavity, including hepatic flexure, splenic flexure and diaphragmatic muscle; and can also improve the accuracy of peritoneal lavage examinations while avoiding blood contamination. Laparoscopic surgery is also a very accurate staging procedure, with potentially reduced complications, bleeding, hospitalization days and expense, and recovery time compared with laparotomy-thus shortening the interval between surgery and initiation of postoperative adjuvant chemotherapy.

However, although some studies have compared laparoscopy and laparotomy for ovarian cancer, most are individual or small-sample case report or case-control studies. A prospective randomized controlled clinical trial is needed.

This will be a prospective, open, parallel, randomized, controlled clinical trial, designed to compare the advantages and disadvantages of laparoscopy and laparotomy in diagnosing and treating early malignant ovarian cancer in terms of surgical safety, postoperative survival rate, reoperation rate, postoperative quality of life and medical cost, to provide evidence for clinical application of laparoscopic surgical staging in in diagnosing and treating early malignant ovarian cancer, and to fill some gaps in the evidence for laparoscopy versus laparotomy. Endoscopic surgical staging of early malignant ovarian cancer accords with the trend of minimal invasion and radical treatment for tumors.

Surgical procedures Laparoscopy: (1) Pneumoperitoneum will be established for laparoscopy. Ascites or pelvic peritoneal lavage fluid will be used for cytologic examination. (2) Unilateral or bilateral attachments will be resected, placed in specimen bags, and removed, to be pathologically examined as fast-frozen samples. Alternatively, the ovarian artery and vein will be ligated, and attachments on the lesion side will be resected and placed in the specimen bag, which will be tied and placed at right iliac fossa. (3) The uterus will be resected and removed through the vagina with the specimen bag at the right iliac fossa. (4) Pelvic and para-aortic lymph nodes will be resected and separately removed through the vagina. (5) The greater omentum below the transverse colon will be resected and, together with parietal peritoneum at the paracolic sulci and basin side, receive multiple punch biopsies. (6) Removal of vermiform appendix; closure of vaginal stump by vaginal suture and laparoscopic suspension; (7) wound hemostasis, irrigation, and drainage.

Laparotomy: Hysterectomy + oophorotomy + high ligation of ovarian artery and vein + dissection of pelvic and abdominal aortic lymph nodes + resection of greater omentum + resection of vermiform appendix. Procedures are the same as with the laparoscopy group.

Withdrawal process Criteria for withdrawal during the trial Patients may withdraw from the trial (1) if the researchers consider withdrawal to be medically necessary, (2) if patients ask to withdraw, or (3) if patients who have no fixed means of contact plan to move to other cities during follow-up.

Withdrawal of consent during follow-up If patients or their families do not agree to do further tests during follow-up, we will not conduct further evaluation. The corresponding data will not be collected, although data previously collected will be retained, and can be used for analysis with informed consent.

Data archiving, collection and monitoring Paper-based case report forms will be archived, and their data will be converted to an electronic version by professionals using a double-data entry strategy.

To ensure the safety of the patient and the integrity of the clinical data, correct informed consent procedures and assessment of primary end points and compliance will be monitored by professional inspectors. Inspectors have the right to query key documents. Besides site visits, inspectors and the test center will keep in touch through email and phone.

Security of patients' data Each patient will be encoded separately during the trial. Case report forms will be saved in accordance with local data protection laws. These data will be strictly confidential. During clinical interviews, clinical research associates will examine patient-related data to ensure its correctness and completeness, and its preservation in accord with legal requirements.

Statistical analysis Statistical analysis will be performed using Statistical Product and Service Solutions(SPSS) 18.0 software, with normally distributed variables expressed as mean ± standard deviation; abnormally distributed variables as median and interquartile range; and categorical variables expressed as number and percentage. Continuous variables will be compared among groups using Student's t-test. Abnormally distributed data will be compared among groups using non-parametric Mann-Whitney U test. Categorical variables will be compared among groups using Chi-square test or Fisher's exact test. Repeated measure analysis of variance (ANOVA) will be performed for the different time point assessments between groups. P < 0.05 will be considered significant.

Contact and communication Our communication strategy mainly involves patients enrolled in trials, who can consult with doctors, family members or friends to decide whether to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative examination indicates highly suspected early stage of ovarian cancer.
* This is the first time treatment to the patient for the ovarian cancer.
* Family consents are granted.

Exclusion Criteria:

* Pregnancy or breast-feeding women
* History of multiple pelvic surgeries; severe adhesions suspected at the surgical area
* Highly allergic constitution or a history of severe allergies
* Systemic infection or severe local infection
* Age younger than 18 years old or older than 65 years old
* Severe cardiopulmonary disease, liver and kidney dysfunction and other severe underlying disease
* Poor compliance (cannot finish the trial) or the investigator believes that the patient is not appropriate for treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Time to recurrence

SECONDARY OUTCOMES:
Overall survival | 5 years
  Time to last follow up/death
Operative complication rate | 30 days
  Intra- and post-operative complication rate of both group
Quality of life after surgery | Baseline, 1 week, 1 month, 3 months and 1 year after surgery
  Quality of life before surgery, and at 1 week, 1 month, 3 months and 1 year after surgery in both groups will be evaluated using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yang, M.D., Principal Investigator — Shengjing Hospital

IPD SHARING:
Plan to Share IPD: Undecided